CLINICAL TRIAL: NCT02241798
Title: Effects of Pre-oxygenation on Indicators of Gas Exchange and Autonomic Function During Seizures in the Epilepsy Unit
Brief Title: Pre-oxygenation and Measures of Gas Exchanges During Seizures in the Epilepsy Monitoring Unit
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator is leaving the institution and has terminated the study.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S13-00435
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Epilepsy
Keywords: epilepsy; oxygen saturation; transcutaneous carbon dioxide; sudep; pre-oxygenation
MeSH Terms: conditions — Epilepsy; Sudden Unexpected Death in Epilepsy | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-oxygenation first (Experimental): 1. st, 3rd, 5th, etc seizure: continuous 'pre-oxygenation' up to 4L O2 nasal prongs, as tolerated
  2. nd, 4th, 6th, etc seizure: Standard practice (O2 only in post-ictal period).
  Interventions: Other: oxygen
- Standard practice first (Experimental): 1. st, 3rd, 5th, etc seizure: Standard practice (O2 only in post-ictal period).
  2. nd, 4th, 6th, etc seizure: continuous 'pre-oxygenation' up to 4L O2 nasal prongs, as tolerated
  Interventions: Other: oxygen

INTERVENTIONS:
Other: oxygen — O2 by nasal prongs

SUMMARY:
The primary goal of the study is to assess the effect of pre-oxygenation on oxygen and carbon dioxide levels during seizures in patients admitted at the Epilepsy Monitoring Unit (EMU). The investigators hypothesize that providing oxygen prior to seizures will help eliminate the drops in changes seen during seizures, such as the drop in oxygen saturation and increase in carbon dioxide levels.

Research will be done on patients that are admitted to the EMU specifically to have seizures occur and to be recorded on video electroencephalography (vEEG), and the only research intervention will be the use of oxygen prior to some of the seizures.

The importance of this research relates to the phenomenon of sudden unexplained death in epilepsy patients (SUDEP). SUDEP cases are typically patients with epilepsy who are found dead by their families in the morning, without a clear cause for death. The risk of SUDEP is as high as 9.3 per 1000 person-years (Shorvon and Tomson 2011). There may be multiple mechanisms for SUDEP to occur, however a leading hypothesis is a decrease in ventilation during the seizure leading to hypoxia. Blood oxygen saturation levels have been found to decrease significantly in 25-50% of patients during or shortly after a seizure while being monitored in hospitals. In rare situations, a significantly lowered oxygen level may trigger a cascade of events from which the body may not be able to recover, leading to SUDEP. In animal models, providing oxygen prior to seizures occurring has been shown to eliminate oxygen desaturation, but more importantly eliminate mortality in animals prone to death due to seizures.

Pre-oxygenation is a standard procedure during rapid-sequence induction anesthesia as it reduces the risk of oxygen desaturation during the apneic period of the procedure. On room air, the estimated duration of safe apnea is 1 minute, but this can increase to 8 minutes following pre-treatment with high FiO2 (Weingart and Levitan 2012). This is primarily due to oxygen replacing nitrogen within alveoli, creating a reservoir of oxygen within the lungs from which transfer to the bloodstream can continue despite the lack of ventilation. The apneic episode during seizures should benefit from the same principle.

The main purpose of the Epilepsy Monitoring Unit (EMU) is to evaluate patients to better characterize seizures, to identify the main seizure focus. In addition to standard EEG with electrodes on the scalp, some patients require invasive localization of the epileptic focus by surgically placing electrodes within the skull (often referred to as GRID patients) on or within the brain, with the goal of being able to resect the area that is causing seizures. To identify where seizure originate electrically, it requires that seizures occur during the vEEG procedure. To provoke seizures, medications are typically lowered, and both partial seizures and those with secondary generalization to full tonic-clonic (GTC) seizures will occur. Prior research has shows that oxygen desaturation below 90% occurs with some complex partial seizures, but hypoxia is more common and more profound with GTCs. Some centers use oxygen saturation and CO2 monitors as their standard of care, and at NYULMC the investigators also have the capability for both for clinical usage.

Oxygen is not currently a mandated standard-of-care, but is often provided by nasal prongs following seizures as part of the post-ictal nursing care, though there is no outcome data to support its use. It is unknown whether pre-treatment with oxygen will reduce the rate of oxygen desaturations clinically, as seen in animal models, and this is the goal of this research project.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-70 yo admitted for monitoring and capturing seizures at the EMU with scalp electrodes and for seizure localization with implantation of intracranial electrodes.

Exclusion Criteria:

* patients who are considered healthy enough to provoke seizure activity will have few medical illnesses severe enough to be of concern with respect to continuous oxygen delivery. However, patients will be screened for moderate to severe chronic obstructive pulmonary disease and excluded, as their minute ventilation may decrease and CO2 levels increased with continuous oxygen supplementation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Oxygen desaturation below 92% following GTCs | during and up to 6 minutes following the seizure

SECONDARY OUTCOMES:
Oxygen Desaturations below 80% following GTCs | during and up to 6 minutes following seizures

CONTACTS AND LOCATIONS:
Locations (1):
- NYU Langone Medical Center, New York, New York, United States